CLINICAL TRIAL: NCT00593671
Title: Preimplantation Genetic Screening for Aneuploidy in Embryos After in Vitro Fertilization in Women Over 35: a Prospective Controlled Randomized Study.
Brief Title: Preimplantation Genetic Screening in Women Over 35 Year
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Thomas D'Hooghe, Leuven University Fertility Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: sdbroc0
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: In Vitro Fertilization
Keywords: aneuploidies in 7 chromosomes increased with advanced maternal age

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PGS group (Active Comparator)
  Interventions: Procedure: Preimplantation genetic screening after embryo biopsy
- control group (No Intervention)

INTERVENTIONS:
Procedure: Preimplantation genetic screening after embryo biopsy — Preimplantation genetic screening after embryo biopsy
  Arms: PGS group

SUMMARY:
In view of insufficient evidence to routinely use Preimplantation Genetic Screening (PGS) to improve success rates after IVF, we test the hypothesis that patients with advanced maternal age (AMA) have a higher implantation rate (IR) after embryo transfer (ET) of chromosomally normal embryos following PGS compared to patients who had an ET without PGS.

In a randomized controlled trial (RCT) in patients with AMA (≥ 35 years), the clinical IR per embryo transferred will be compared after ET on day 5 or 6 between the PGS group (embryo biopsy and analysis of chromosomes 13, 16, 18, 21, 22, X and Y) and the control group without PGS.

ELIGIBILITY:
Inclusion Criteria:

* All couples with a medical indication for IVF and with a female age of at least 35 years are invited to participate in the study.

Exclusion Criteria:

* Cycles were excluded from the study if ≤ 2 fertilized oocytes were available on day 1 after oocyte retrieval (OR), or if ≤ 2 ≥ 6c stage embryos were available on day 3 after OR.

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2002-06; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Clinical implantation rate per embryo transferred | end of study

SECONDARY OUTCOMES:
Pregnancy rate per transfer | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M D'Hooghe, MD, Study Director — UZ Leuven
Locations (1):
- Leuven University Fertility Center, Leuven, Belgium